CLINICAL TRIAL: NCT01472601
Title: A Prospective Study of Pharmacogenetic Factors and Gene Expression Profile in Patients Receiving Adjuvant Therapy With FOLFOX-6 After Curative Resection of Colon Cancer
Brief Title: A Prospective Study of Pharmacogenetic Factors and Gene Expression Profile
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Suk Park, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2011-04-098
Record Dates: First submitted 2011-11-13; First posted 2011-11-16 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FOLFOX_6: Oxaliplatin : 85 mg/m2/day D1 Leucovorin : 200 mg/m2/day D1 5-FU : 400 mg/m2/day D1 5-FU : 2,400 mg/m2/day D1 over 46 hrs Every 2 weeks, first 6 cycles, then Leucovorin : 200 mg/m2/day D1 5-FU : 400 mg/m2/day D1 5-FU : 2,400 mg/m2/day D1 over 46 hrs Every 2 weeks, 6 cycles
- FOLFOX_12: Oxaliplatin : 85 mg/m2/day D1 Leucovorin : 200 mg/m2/day D1 5-FU : 400 mg/m2/day D1 5-FU : 2,400 mg/m2/day D1 over 46 hrs Every 2 weeks, total of 12 cycles

SUMMARY:
This study is a parallel translational study of a Randomized Phase III trial Investigating the Role of Oxaliplatin duration (6 Cycles Versus 12 Cycles) in modified FOLFOX-6 Regimen as Adjuvant Therapy for Patients with Stage II/III Colon Cancer (MIDAS trial: protocol NCCCTS-467) . Patients participating in the trial will be provided with the informed consent of this parallel study, and peripheral blood and tumor tissue of those who signed the consent will be collected for germline polymorphism analysis and gene expression profile study .

ELIGIBILITY:
Inclusion Criteria:

* Curatively resected, histologically confirmed colon adenocarcinoma (presence of the inferior pole of the tumor above the peritoneal reflection)
* AJCC/UICC high-risk stage II, stage III colon cancer Stage II patient with high risk of relapse, if they fulfill one or more of the following criteria:(T4 tumors,bowel obstruction or perforation,vascular or lymphatic or perineural invasion)
* Patients who are participating in the randomized phase II trial of FOLFOX 6 or 12 cycles
* Patients should sign a written informed consent for this translational study before or during participating in a randomized phase III study investigating the role of oxaliplatin duration (6 cycles versus 12 cycles) in modified FOLFOX-6 regimen as adjuvant therapy for patients with stage II/III colon cancer

Exclusion Criteria:

* Patients who do not agree with sampling of peripheral blood for genetic analysis
* Patients who are considered not to be suitable for this study at investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients should sign a written informed consent for this translational study before or during participating in a randomized phase III study investigating the role of oxaliplatin duration (6 cycles versus 12 cycles) in modified FOLFOX-6 regimen as adjuvant therapy for patients with stage II/III colon cancer
Sampling Method: Probability Sample
Enrollment: 2660 (Estimated)
Dates: Start 2011-05-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 6years
  To estimate the interaction between disease-free survival, duration of adjuvant oxaliplatin treatment, and genotypes concerning DNA repair (ERCC1, XPD, XRCC1) and detoxification (GSTP1)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical Center, Seoul, South Korea